CLINICAL TRIAL: NCT01733420
Title: The Clinical and Radiographic Efficacy of Biodentine™ and White Mineral Trioxide Aggregate in Deciduous Molar Pulpotomy - a Randomized Control Trial
Brief Title: Biodentine Versus White MTA Pulpotomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/538
Record Dates: First submitted 2012-11-07; First posted 2012-11-27 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Extensive Decay in Primary Molars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biodentine (Experimental): Pulpotomy using Biodentine as pulpotomy medicine.
  Interventions: Drug: Biodentine pulpotomy
- White Mineral trioxide Aggregate (MTA) (Active Comparator): Pulpotomy using white MTA as pulpotomy medicine.
  Interventions: Drug: White MTA pulpotomy
- Tempophore (Active Comparator): Pulpotomy using Tempophore as pulpotomy medicine in a control group.
  Interventions: Drug: Tempophore pulpotomy

INTERVENTIONS:
Drug: Biodentine pulpotomy
  Arms: Biodentine
Drug: White MTA pulpotomy
  Arms: White Mineral trioxide Aggregate (MTA)
Drug: Tempophore pulpotomy
  Arms: Tempophore

SUMMARY:
A clinical trial to evaluate and compare three different products used for endodontic treatment (taking the infected nerve out of the teeth) of primary teeth.

Null Hypothesis: The new biological products (WMTA and Biodentine) behave as good as the former iodoform product.

ELIGIBILITY:
Inclusion Criteria:

* Patients (Children with carious deciduous molars indicated for pulpotomy) belonging to the category of ASA I according to the 'American Society of Anaesthesiologists'.
* Patients without any known medical history of systemic complications contradicting pulp treatment.
* Patients are indicated for treatment under general anaesthesia due to polycaries / fear / anxiety / very young age.
* Written consent is obtained from the parent/guardian after explaining the full details of the treatment procedure and its possible outcomes.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2011-10-04 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Clinical successes after pulpotomy. | at baseline visit
  clinical evaluation and radiography of the tooth is performed. Clinical criteria: abscence of post-operative pain, absence of pain on percussion and palpation, absence of abscess or swelling, absence of sinus tract or fistula and absence of pathologic tooth mobility.
Clinical success after pulpotomy. | 3 months after pulpotomy.
  clinical evaluation and radiography of the tooth is performed. Clinical criteria: abscence of post-operative pain, absence of pain on percussion and palpation, absence of abscess or swelling, absence of sinus tract or fistula and absence of pathologic tooth mobility.
Clinical successes after pulpotomy. | 6 months after pulpotomy.
  Clinical evaluation and radiography of the tooth is performed. Clinical criteria: abscence of post-operative pain, absence of pain on percussion and palpation, absence of abscess or swelling, absence of sinus tract or fistula and absence of pathologic tooth mobility.
Clinical successes after pulpotomy. | 12 months after pulpotomy.
  Clinical evaluation and radiography of the tooth is performed. Clinical criteria: abscence of post-operative pain, absence of pain on percussion and palpation, absence of abscess or swelling, absence of sinus tract or fistula and absence of pathologic tooth mobility.
Radiographic successes after pulpotomy. | at baseline visit
  Radiographic criteria: presence of normal periodontal ligament space, absence of internal or external root resorption, absence of canal calcification, absence of periradicular radiolucency and no loss or break of lamina dura.
Radiographic successes after pulpotomy. | 6 months after pulpotomy.
  Radiographic criteria: presence of normal periodontal ligament space, absence of internal or external root resorption, absence of canal calcification, absence of periradicular radiolucency and no loss or break of lamina dura.
Radiographic successes after pulpotomy. | 12 months after pulpotomy.
  Radiographic criteria: presence of normal periodontal ligament space, absence of internal or external root resorption, absence of canal calcification, absence of periradicular radiolucency and no loss or break of lamina dura.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Martens, PhD, DDS, Principal Investigator — University Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium